CLINICAL TRIAL: NCT04532216
Title: The Clinical and Biomechanical Research of the New Arthroscopic Technique for the Treatment of High-grade Dislocation of the Acromioclavicular Joint
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Beijing Jishuitan Hospital (Other)
Responsible Party: Principal Investigator, Chunyan Jiang, Director of Sports Medicine Service of Beijing Jishuitan hospital, Beijing Jishuitan Hospital
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CJiang
Record Dates: First submitted 2020-08-26; First posted 2020-08-31 (Actual); Last update posted 2020-08-31 (Actual); Status verified 2020-08

CONDITIONS: Dislocation of the Acromioclavicular Joint

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Study group (Experimental)
  Interventions: Procedure: Arthroscopic-Assisted Acromioclavicular Joint Reconstruction Using the TightRope Device
- Control group (Other)
  Interventions: Procedure: Traditional surgery

INTERVENTIONS:
Procedure: Arthroscopic-Assisted Acromioclavicular Joint Reconstruction Using the TightRope Device — Arthroscopic-assisted AC joint reconstruction with the TightRope device with allograft augmentation and with the patient in the lateral decubitus position is a method of restoring joint stability
  Arms: Study group
Procedure: Traditional surgery — Tendon transfer
  Arms: Control group

SUMMARY:
Acromioclavicular joint dislocation is a common disease in shoulder surgery, which mostly occurs in young and middle-aged patients. Severe acromioclavicular joint dislocations of Rockwood type IV, V, and VI require surgical treatment. Among them, the common clinical type IV and type V severe acromioclavicular joint dislocations are often treated with autologous/allogenous tendon transplantation and coracoclavicular ligament reconstruction under shoulder arthroscopy. Although this minimally invasive surgical method has certain advantages over incision surgery, due to factors such as poor healing after tendon transplantation and failure of coracoclavicular fixation, the recurrence rate of postoperative dislocation is still as high as 30%, which seriously affects the prognosis of patients. Therefore, we proposed a new surgical technique of minimally invasive shoulder arthroscopic coracoclavicular suspension fixation and coracoclavicular ligament residual reconstruction, which aims to strengthen the fixation strength of the coracoclavicular space, promote the healing of the coracoclavicular ligament, and reduce the recurrence rate of postoperative dislocation. To improve postoperative shoulder joint function of patients. This project intends to use non-randomized controlled clinical research and biomechanical research to compare traditional surgical techniques with new microscopic techniques in terms of surgical efficacy, postoperative complications, and internal plant fixation strength to establish the therapeutic advantages of the new technology. Its application and promotion provide important clinical evidence to improve the treatment of severe acromioclavicular joint dislocation in the field of shoulder surgery.

ELIGIBILITY:
Inclusion Criteria:

* Consecutive cases of coracoclavicular ligament reconstruction surgery usingTightRope Device With Allograft Augmentation and shoulder arthroscopic reconstruction of coracoclavicular ligament with autologous/allogeneic tendon transplantation.
* Injury type Rockwood type IV and V type severe acromioclavicular joint dislocation
* The time from injury to operation is less than 3 weeks

Exclusion Criteria:

* Combined with neurovascular injury
* Previous history of ipsilateral shoulder surgery
* The patient refused to sign the informed consent and participate in the trial

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 54 (Estimated)
Dates: Start 2020-09-01 (Estimated); Primary Completion 2022-06-30 (Estimated); Study Completion 2023-06-30 (Estimated)

PRIMARY OUTCOMES:
ASES score | 1 year postoperatively
  The ASES score is a 10-item measure of shoulder pain and function

CONTACTS AND LOCATIONS:
Overall Officials: Chunyan Jiang, Study Chair — Sports Medicine Service, Beijing Jishuitan hospital

IPD SHARING:
Plan to Share IPD: Undecided